CLINICAL TRIAL: NCT06730269
Title: Comparative Efficacy of Face-to-Face and Telerehabilitation Approaches in Managing Thoracic Hyperkyphosis Among 9-12-Year-Olds: a Randomized Clinical Trial
Brief Title: Face-to-Face Vs. Telerehabilitation for Thoracic Hyperkyphosis in Children: a Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Seda GÖZENER CANBÜLBÜL, PhD candidate, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: İMU-SEDAGOZENER-004
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Kyphosis Thoracic; Hyperkyphosis
Keywords: Thoracic hyperkyphosis; face-to-face rehabilitation; telerehabilitation; spinal posture; musculoskeletal health; corrective exercises; Pediatric Kyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Face-to-Face Rehabilitation Group (Experimental): Participants in this arm received a thoracic corrective exercise program in person, consisting of four exercises targeting back extensor muscles. The exercises were performed three times a week for six weeks under the supervision of a trained therapist.
  Interventions: Behavioral: Face-to-Face Rehabilitation Program
- Telerehabilitation Group (Experimental): Participants in this arm followed the same thoracic corrective exercise program, but the sessions were delivered online through the Fiziu platform. Exercises were performed three times a week for six weeks with remote guidance and monitoring.
  Interventions: Behavioral: Telerehabilitation Program

INTERVENTIONS:
Behavioral: Face-to-Face Rehabilitation Program — The Face-to-Face Rehabilitation Program is a structured rehabilitation regimen designed to improve posture, reduce pain, and strengthen back extensor muscles in children with thoracic hyperkyphosis. Participants in this group engaged in the Thoracic Corrective Exercise Program, which included four specific exercises targeting thoracic spine correction. The exercises were performed three times per week over six weeks, under the direct supervision of a trained therapist. This setup ensured real-time feedback, personalized adjustments, and guidance during each session, optimizing the effectiveness of the rehabilitation process.
  Arms: Face-to-Face Rehabilitation Group
Behavioral: Telerehabilitation Program — The Telerehabilitation Program is a structured rehabilitation regimen designed to improve posture, reduce pain, and strengthen back extensor muscles in children with thoracic hyperkyphosis. Participants in this group followed the Thoracic Corrective Exercise Program, which included four specific exercises targeting thoracic spine correction, performed three times per week over six weeks. The program was delivered remotely through the Fiziu platform, allowing therapists to provide virtual guidance, feedback, and monitoring during the sessions. This approach offered flexibility for families and ensured accessibility to rehabilitation services from the comfort of their homes.
  Other Names: Fiziu Platform Video Based Exercise Group
  Arms: Telerehabilitation Group

SUMMARY:
This study evaluates the effectiveness of face-to-face versus telerehabilitation programs for children aged 9-12 with thoracic hyperkyphosis, a condition caused by poor posture that leads to excessive forward curvature of the spine. Twenty children participated in a six-week corrective exercise program, either in person or through an online platform. Both approaches significantly improved spinal posture, back muscle strength, and pain levels, with no notable differences in outcomes between the two methods. The findings suggest that telerehabilitation is as effective as face-to-face rehabilitation, offering a flexible option for managing thoracic hyperkyphosis in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9-12 years.
* Diagnosed with thoracic hyperkyphosis (Thoracic Kyphosis Angle > 40 degrees).
* Able to participate in a 6-week rehabilitation program (face-to-face or telerehabilitation).

Exclusion Criteria:

* Children with congenital spinal malformations.
* Children with mental health issues that could interfere with participation or compliance in the study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Thoracic Kyphosis Angle (TKA) | 6 weeks
  It was measured using a flexicurve ruler to assess the curvature of the thoracic spine before and after the intervention.
  >45° is considered hyperkyphosis
Manual Muscle Test (MMT) | 6 weeks
  Evaluates back muscle strength before and after the intervention. Minimum = 0 (no muscle contraction), Maximum = 5 (normal muscle strength).
Visual Analog Scale (VAS) | 6 weeks
  Assesses pain levels before and after the intervention. Minimum = 0 (no pain), Maximum = 10 (worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Seda Gözener Canbülbül, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Kavacık, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang L, Lu X, Yan B, Huang Y. Prevalence of Incorrect Posture among Children and Adolescents: Finding from a Large Population-Based Study in China. iScience. 2020 May 22;23(5):101043. doi: 10.1016/j.isci.2020.101043. Epub 2020 Apr 8. PMID 32330860
- [Background] Feng Q, Wang M, Zhang Y, Zhou Y. The effect of a corrective functional exercise program on postural thoracic kyphosis in teenagers: a randomized controlled trial. Clin Rehabil. 2018 Jan;32(1):48-56. doi: 10.1177/0269215517714591. Epub 2017 Jun 14. PMID 28610442
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28610442/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32330860/